CLINICAL TRIAL: NCT03707834
Title: Partnering With WIC to Prevent Excessive Weight Gain in Pregnancy
Acronym: GWG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25256; R01DK115939-01A1 (NIH)
Record Dates: First submitted 2018-09-13; First posted 2018-10-16 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight; Pregnancy Related
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WIC Standard Care (SC) (No Intervention): Participants assigned to the WIC standard care arm will receive usual care offered to pregnant women at WIC.
- Antenatal Obesity Treatment (AO) (Experimental): The AO arm consists of a multi-component, theory- and evidence-based intervention and includes weight-related behavior change through goal setting and self-monitoring, behavioral skills training, interpersonal support, and social modeling strategies.
  Interventions: Behavioral: Antenatal Obesity Treatment (AO)

INTERVENTIONS:
Behavioral: Antenatal Obesity Treatment (AO) — Participants in the treatment (AO) arm will receive a 4-component intervention: 1)Behavior change goals; 2)Self-monitoring; 3)Tailored skills training; and 4)WIC provider counseling Both treatment and usual care arms will receive the current standard of care offered to postpartum mothers at WIC.
  Arms: Antenatal Obesity Treatment (AO)

SUMMARY:
The purpose of this study is to determine the effect of an antenatal obesity treatment on gestational weight gain when integrated into Philadelphia WIC.

DETAILED DESCRIPTION:
Institute of Medicine (IOM) guidelines for weight gain in pregnancy are clear, but evidence-based treatment approaches are not widely available. This evidence gap is particularly pressing for medically vulnerable women - those who are low income and often racial/ethnic minorities. These women have the highest rates of obesity, but almost no resources to support weight control in pregnancy. Without intervention, most will exceed Institute of Medicine recommended gains and incur significant morbidity for themselves and their children. There is preliminary data from the investigators supporting the efficacy of digital health platforms for delivering antenatal obesity treatment among the medically vulnerable. However, the investigators' inexpensive, easily scalable approach has not been integrated and tested in real world settings, limiting broad reach and dissemination potential. Dissemination considerations are especially pressing for socioeconomically disadvantaged and minority populations because of these groups' higher obesity risk, greater potential for experiencing obesity-related comorbidities in pregnancy, and limited finances to afford alternative treatments. The Women, Infants and Children (WIC) Food and Nutrition Program is the leading public health nutrition program for pregnant women and their children in the US, and thus, it is in a unique position to meaningfully impact the obesity epidemic among the more than 9 million disadvantaged participants it serves annually. Yet no demonstrations of effective gestational weight gain interventions exist in WIC. The investigators propose a pragmatic trial designed to rigorously test their antenatal obesity treatment approach integrated into Philadelphia WIC community clinics. The investigators have long-standing relationships with WIC staff and prior experience conducting pragmatic clinical trials in under-resourced settings. The investigators will randomize 438 African American and Hispanic Philadelphia County WIC participants with obesity in early pregnancy to one of two treatment arms: 1) standard WIC care; or 2) an antenatal obesity treatment arm, which includes empirically supported behavior change goals, regular self-monitoring text messages with automated feedback, tailored skills training materials, and counseling from WIC nutritionists. The primary outcome is prevalence of excessive gestational weight gain; the investigators will additionally examine changes in diet and physical activity, health-related quality of life, and rates of adverse pregnancy outcomes. They will use the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework to evaluate the intervention's dissemination potential and cost effectiveness in the WIC setting. The proposed project will constitute the first systematic translation of a comprehensive antenatal obesity treatment program focused on low-income, racial/ethnic minorities, using the strengths of mHealth (mobile health) and WIC provider counseling for intervention delivery.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 kg/m2
* Self-identify as African American or Hispanic
* Gestational age ≤16 weeks' (measured using last menstrual period)
* Philadelphia WIC participant
* Willingness to receive study texts
* Own a cell phone with an unlimited text messaging plan
* Able to participate in light to moderate physical activity (walking)

Exclusion Criteria:

* Prior bariatric surgery
* Pre-existing medical condition that could influence weight (e.g., diabetes, HIV, thyroid disorder, bulimia, anorexia, gallbladder disease)
* Diagnosis contraindicating weight control (e.g., hyperemesis gravidarum)
* Shared phone
* Multiple pregnancy (e.g., twins)
* Current and/or previous participant for our Temple-led obesity treatment interventions in pregnancy or the postpartum period
* Serious or unstable medical or psychological conditions that, in the opinion of the PI, would compromise the subject's safety for successful participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon J Herring, MD, MPH, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Dr. Herring (PI) will ensure that all publications that result from data collected as part of this project will comply with the NIH public access policy. Also, Dr. Herring agrees to develop a transportable de-identified database, codebook, and mechanism by which data can be shared with other investigators upon approval of the study's research team. The Resource Sharing Plan will be reviewed and approved by Temple University's Institutional Review Board.

RESULTS

PARTICIPANT FLOW:
Groups:
- Antenatal Obesity Treatment (AO): The AO arm consists of a multi-component, theory- and evidence-based intervention and includes weight-related behavior change through goal setting and self-monitoring, behavioral skills training, interpersonal support, and social modeling strategies.
  Antenatal Obesity Treatment (AO): Participants in the treatment (AO) arm will receive a 4-component intervention: 1)Behavior change goals; 2)Self-monitoring; 3)Tailored skills training; and 4)WIC provider counseling
  Both treatment and usual care arms will receive the current standard of care offered to postpartum mothers at WIC.
Period: Overall Study
Arm/Group | WIC Standard Care (SC) | Antenatal Obesity Treatment (AO)
Started | 207 | 209
Completed | 196 | 197
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Population: Baseline analyses include all participants randomized whether or not they competed the study. 416 participants were randomized even though only 393 participants completed the study and were included in the primary outcomes analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | WIC Standard Care (SC) | Antenatal Obesity Treatment (AO) | Total
Number analyzed (Participants) | 207 | 209 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (5.6) | 29.2 (5.6) | 29.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 209 | 416
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 66 | 136
  Not Hispanic or Latino | 137 | 143 | 280
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 144 | 148 | 292
  White | 3 | 5 | 8
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 59 | 56 | 115
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 207 | 209 | 416
BMI, Categorical: 25-29.9 kg/m^2 (with overweight); >=30 kg/m2 (with obesity) [Count of Participants; unit: Participants]
  BMI >=30 kg/m^2 (with obesity) | 155 | 152 | 307
  BMI 25-29.9 kg/m^2 (with overweight) | 52 | 57 | 109
Parity: Nulliparous, Primi- & Multiparous [Count of Participants; unit: Participants]
  Nulliparous | 53 | 74 | 127
  Primi- & Multiparous | 154 | 135 | 289
Education: More than High School, High School and Below [Count of Participants; unit: Participants]
  More than High School | 95 | 98 | 193
  High School and Below | 112 | 111 | 223
Gestational Age, Continuous [Mean (Standard Deviation); unit: weeks] | 15.4 (2.5) | 15.4 (2.4) | 15.4 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women With Excessive Gestational Weight Gain
Description: Excessive weight gain is defined as the percentage of mothers exceeding weekly IOM weight gain targets (>0.32 kg/week for BMI 25-29.9 kg/m2; >0.27 kg/week for BMI ≥30 kg/m2) over the study period (from enrollment to end of pregnancy).
Time Frame: End of Pregnancy (36-38 weeks' gestation)
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Standard Care (SC) | Antenatal Obesity Treatment (AO)
Number analyzed (Participants) | 196 | 197
Participants | 126 | 119

2. Primary Outcome: Change in Maternal Weight
Description: Weight gain will be calculated as the difference between weight in kilograms measured at 36-38 weeks' gestation and baseline weight.
Time Frame: At baseline (<16 weeks' gestation) and End of Pregnancy (36-38 weeks' gestation)
Measure: Median (Inter-Quartile Range); unit: kilograms
Arm/Group | WIC Standard Care (SC) | Antenatal Obesity Treatment (AO)
Number analyzed (Participants) | 196 | 197
kilograms | 7.6 [4.0 to 11.5] | 7.2 [4.0 to 11.4]

3. Secondary Outcome: Change in Dietary Intake
Description: Will be measured using the Automated Self-Administered 24-hour (ASA24) dietary assessment tool, a web application developed by NCI. We will collect 3 separate 24-hour dietary recalls (1 weekend day, 2 weekdays) at baseline and 36-38 weeks' gestation.
Time Frame: Baseline and 36-38 weeks' gestation
Reporting Status: Not Posted, anticipated posting 2026-06

4. Secondary Outcome: Percentage With Glucose Intolerance
Description: Evaluated via medical record abstraction
Time Frame: Delivery
Reporting Status: Not Posted, anticipated posting 2026-06

5. Secondary Outcome: Percentage With Hypertension
Description: Evaluated via medical record abstraction
Time Frame: Delivery
Reporting Status: Not Posted, anticipated posting 2026-06

6. Secondary Outcome: Change in Maternal 6-month Weight Postpartum (pp)
Description: Weight change will be calculated as the difference between mean 6-month PP weight and baseline weight in kilograms.
Time Frame: At baseline and 6-month PP
Reporting Status: Not Posted, anticipated posting 2026-06

7. Secondary Outcome: Change in Maternal 12-month Weight Postpartum (pp)
Description: Weight change will be calculated as the difference between mean 12-month PP weight and baseline weight in kilograms.
Time Frame: At baseline and 12-month PP
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline/enrollment through end of pregnancy, up to 26 weeks total (primary outcome data collection period).
Arm/Group | WIC Standard Care (SC) | Antenatal Obesity Treatment (AO)
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/209
Serious Adverse Events (participants affected / at risk) | 0/207 | 0/209
Other Adverse Events (participants affected / at risk) | 0/207 | 0/209

LIMITATIONS AND CAVEATS:
Findings need to be considered in light of the Covid-19 pandemic, which led to challenges with intervention delivery and intensity (i.e., limited in-person WIC visits, structural impediments for system-wide adaptation) along with remote weight and height measures for some participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03707834/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT03707834/ICF_001.pdf